CLINICAL TRIAL: NCT06683157
Title: Natural History of Isolated Calf Vein Thrombosis - A Prospective Cohort Under Ultrasound Surveillance
Status: Recruiting | Type: Observational
Sponsor: Stadtisches Klinikum Dresden (Other)
Responsible Party: Principal Investigator, Kerstin Spranger, Prof. Dr. med. S.M. Schellong, Stadtisches Klinikum Dresden
Other Study IDs: ICVT
Record Dates: First submitted 2024-10-17; First posted 2024-11-12 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Acute Embolism and Thrombosis of Calf Muscular Vein
Keywords: Isolated Calf Vein Thrombosis; ultrasound surveillance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- serial ultrasound 3: CCUS will be repeated on day 5±2 , day 10±2 and day 30±4. If the ICVT has propagated into the trifurcation area, the popliteal vein, or into more proximal veins therapy will be implemented according to current guidelines for proximal DVT. If no propagation to proximal veins has occurred anticoagulation will be withheld further on.
  Interventions: Diagnostic Test: not drug

INTERVENTIONS:
Diagnostic Test: not drug — Patients presenting with symptomatic ICVT will be examined by CCUS for both legs. Inclusion/exclusion criteria will be checked. No anticoagulation therapy is given. Compression stockings at the calf length will be prescribed for 30 days.
  CCUS will be repeated on day 5±2, day 10±2, and day 30±4. If the ICVT has propagated into the trifurcation area, the popliteal vein, or into more proximal veins therapy will be implemented according to current guidelines for proximal DVT. If no propagation to proximal veins has occurred anticoagulation will be withheld further on.
  Other Names: ultrasound surveillance

SUMMARY:
The treatment of ICVT is still controversial as conflicting international guideline strategies show. Evidence suggests that propagation rates of ICVT without risk factors are low. Unless ICVT propagates to proximal veins anticoagulation can safely been withheld, thereby avoiding a bleeding risk for the patient. However, the impact of different risk factors on propagation rates is not well understood. This gap in knowledge can only be filled by a natural history study of ICVT without anticoagulation. Since patients are safe as long as no propagation occurs close ultrasound surveillance is an adequate safety umbrella for the natural history study period. In addition, it provides an objective outcome measure to define the impact of risk factors.

DETAILED DESCRIPTION:
For the purpose of this study, ICVT is defined as any thrombus being present in the calf muscle veins and/or in the deep paired calf veins as long as they do not affect the confluence (trifurcation) area or the popliteal vein.

Patients presenting with symptomatic ICVT will be examined by CCUS for both legs (V1). Inclusion/exclusion criteria will be checked, and patients will be informed about the nature of the study. In case patients provide informed consent, no anticoagulation therapy is given. Compression stockings at the calf length will be prescribed for 30 days.

CCUS will be repeated on day 5±2 (V2), day 10±2 (V3), and day 30±4 (V4). If the ICVT has propagated into the trifurcation area, the popliteal vein, or into more proximal veins therapy will be implemented according to current guidelines for proximal DVT. If no propagation to proximal veins has occurred anticoagulation will be withheld further on

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptomatic ICVT proven by CCUS
* Absence of proximal DVT or PE
* Age of 18 or older
* Outpatient and inpatient status
* Written informed consent

Exclusion Criteria:

* Bedridden patients
* Prior unprovoked VTE
* Active malignancy (diagnosis within the last 6 months, and/or incomplete resection, and/or ongoing radiotherapy or chemotherapy, and/or metastatic disease).
* Pregnancy
* Therapeutic anticoagulation therapy for reasons other than VTE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with symptomatic ICVT will be examined by CCUS for both legs. Inclusion/exclusion criteria will be checked. No anticoagulation therapy is given.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-09-18 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of proximal extension of DVT and / or pulmonary embolism, symptomatic or asymptomatic DVT | Day 30
  Proximal DVT has to be documented by CCUS as a new thrombus in the trifurcation area, the popliteal vein, or in more proximal deep veins. Non-fatal PE has to be documented as an intraluminal filling defect in CT pulmonary angiography, as an unequivocal perfusion defect in lung scintigraphy, preferably performed in SPECT technique, or, in case of hemodynamic compromise, by echocardiographic signs of right ventricular failure and/or direct thrombus visualization.

CONTACTS AND LOCATIONS:
Locations (1):
- Städtisches Klinikum Dresden, Dresden, Saxony, Germany